CLINICAL TRIAL: NCT02265939
Title: Phase Ⅱ Dose Response Study of NPO-13 in Patients Undergoing Total Colonoscopy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Nihon Pharmaceutical Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Diagnostic
Other Study IDs: NPO-13
Record Dates: First submitted 2014-10-11; First posted 2014-10-16 (Estimated); Last update posted 2021-11-16 (Actual); Status verified 2015-04

CONDITIONS: Bowel Disease
MeSH Terms: conditions — Intestinal Diseases

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- 0% NPO-13 (Placebo Comparator): Placebo
  Interventions: Drug: NPO-13
- 0.2% NPO-13 (Active Comparator): Low dose
  Interventions: Drug: NPO-13
- 0.4% NPO-13 (Active Comparator): Medium dose
  Interventions: Drug: NPO-13
- 0.8% NPO-13 (Active Comparator): High dose
  Interventions: Drug: NPO-13

INTERVENTIONS:
Drug: NPO-13

SUMMARY:
Patients who require screening colonoscopy will receive an intraluminal spraying of NPO-13 per contraction region of large bowel up to fifth times during the colonoscopy.

The efficacy of NPO-13 will be evaluated based on the proportion of the splayed region with no contraction after NPO-13 dosage (primary outcome measure). The colonic spasm will be assessed by an independent committee using recorded video images.

The safety of NPO-13 will be evaluated based on adverse events and adverse drug reactions (ADRs) observed between administration and seven days after administration.

ELIGIBILITY:
Inclusion Criteria:

Inpatients or outpatients of either sex who visit medical institutions for treatment or follow-up of confirmed or suspected colonic disease (symptoms) and meet the criteria (1) and (2) below will be enrolled in the study. Patients have to provide written informed consent for voluntary participation in the study.

1. Patients who need colonoscopy
2. Patients who are older than 20 years at the time of consent

Exclusion Criteria:

1. Patients with a history of abdominal surgical treatment (including the laparoscopic surgery) including the gynecology operation
2. Patients with contraindication to colonoscopy including the paralytic ileus
3. Patients with a history of shock or hypersensitivity to l-menthol or peppermint oil (mint oil)
4. Patient with contraindication to bowel cleansing preparation
5. Patients on cancer treatment (chemotherapy or radiotherapy)
6. Patients who need sedative colonoscopy
7. Patients who receives a therapeutic colonoscopy
8. Pregnant or lactating women, women of childbearing potential, or women who plan to become pregnant during the study
9. Patients who have received other investigational drugs within four months before consent or who are participating in other clinical studies
10. Patients who have been exposed to NPO-13
11. Patients otherwise ineligible for participation in the study in the investigator's or subinvestigator's opinion

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 132 (Actual)
Dates: Start 2014-10; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
The proportion of the splayed region with no contraction after NPO-13 dosage | 3 min

SECONDARY OUTCOMES:
The proportion of the splayed region with an onset of action | 3 min
The proportion of patients with no contraction in all the sprayed regions | 3 min
The proportion of patients with no contraction in one or more the sprayed region | 3 min
Change in colonic contraction | 3 min
Adverse events and ADRs observed between administration and 7 ± 3 days after administration | up to 10 days

CONTACTS AND LOCATIONS:
Locations (3):
- Japan (3):
  - Fukuoka
  - Osaka
  - Tokyo